CLINICAL TRIAL: NCT05708443
Title: Effect of Combined Upper and Lower Extremity Endurance Training Versus Lower Extremity Training Alone on ADL and Walking in COPD Patients
Brief Title: Effect of Combined Endurance Training on ADL and Walking in COPD Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICS Maugeri CE2711
Record Dates: First submitted 2023-01-12; First posted 2023-02-01 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: COPD
Keywords: ADL; COPD; Glittre Test; exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lower limbs (LL) group (Active Comparator): These patients will participate in a pulmonary rehabilitation program (usual training) on lower limbs
  Interventions: Other: LL group
- lower plus upper limbs (L+UL) group (Experimental): These patients will attend a rehabilitation program combining upper and lower extremity training
  Interventions: Other: L+UL group

INTERVENTIONS:
Other: LL group — The program will include daily sessions of 90 minutes, for a total of 14 sessions, consisting of:
  1. 60 minutes on a stationary bike for the lower limbs (2 sessions per day of 30 minutes) at moderate-high intensity;
  2. 30 minutes of strengthening exercises for upper limbs (biceps, pectoral, latissimus dorsi) and lower limbs (quadriceps, gluteus and hamstrings) performed free body or with the aid of weights.
  All sessions will be supervised by a physiotherapist.
  Other Names: Active Comparator
  Arms: lower limbs (LL) group
Other: L+UL group — These patients will attend a rehabilitation program with daily sessions of 90 minutes, for a total of 14 sessions, consisting of:
  1. 30 minutes on a stationary bike for the lower limbs (1 session of 30 minutes per day) at moderate-high intensity;
  2. 30 minutes with arm-ergometer (1 daily session of 30 minutes) at moderate-high intensity;
  3. 30 minutes of strengthening exercises for upper limbs (biceps, pectoral, latissimus dorsi) and lower limbs (quadriceps, gluteus and hamstrings) performed free body or with the aid of weights.
  All sessions will be supervised by a physiotherapist.
  Other Names: Experimental
  Arms: lower plus upper limbs (L+UL) group

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a chronic disease with related exercise intolerance and marked disability due to symptoms such as dyspnea and fatigue. Effort intolerance and exercise-induced symptoms cause marked impairment in completing activities of daily living (ADL). Pulmonary rehabilitation (PR), which has exercise as a major component, is considered a key treatment in the management of COPD since PR is effective in improving exercise tolerance, exercise-induced dyspnea and fatigue, and health-related quality of life. Rehabilitation is also effective in improving the time required to perform ADLs, reducing symptoms and disability. Studies show that rehabilitation protocols with upper limb exercises added to lower limb training are able to give additional benefits in terms of effort tolerance (endurance time at the arm ergometer and oxygen consumption) and reduction of dyspnea at iso-load.

The primary aim of this study is to evaluate whether the combined "arm and leg" training modality, compared to a gold standard protocol -involving only the lower limbs training- is more effective in improving ADL performance in terms of reduction of exercise time for a specific test (GLITTRE test).

DETAILED DESCRIPTION:
Background:

Chronic Obstructive Pulmonary Disease (COPD) is a chronic disease with related exercise intolerance and marked disability due to symptoms such as dyspnea and fatigue. Effort intolerance and exercise-induced symptoms cause marked impairment in completing activities of daily living (ADL). COPD patients often rely on a caregiver to perform some ADLs for intolerable dyspnea and fatigue since the early stages of the disease. In fact, even while performing simple ADLs, COPD patients develop dynamic hyperinflation and reach a ventilatory limit that forces them to stop or slow down. Symptoms and disability worsen the patient's quality of life.

Pulmonary rehabilitation (PR), which has exercise as a major component, is considered a key treatment in the management of COPD since PR is effective in improving exercise tolerance, exercise-induced dyspnea, and fatigue, and health-related quality of life. Rehabilitation is also effective in improving the time required to perform ADLs, reducing symptoms and disability.

Lower extremity cycle ergometer training improves peak oxygen uptake, and reduces heart rate, minute ventilation, dyspnea, and leg fatigue at submaximal work speeds. Moreover, upper limb training has been described to reduce dyspnea, increase respiratory muscle strength, and have an effect on patients' global exercise tolerance.

Studies show that rehabilitation protocols with upper limb exercises added to lower limb training are able to give additional benefits in terms of effort tolerance (endurance time at the arm ergometer and oxygen consumption) and reduction of dyspnea at iso-load.

To our knowledge, no study has investigated training programs in COPD patients with similar timing of intervention comparing selective lower extremity endurance training with combined upper and lower extremity training.

The primary aim of this study is to evaluate whether the combined "arm and leg" training modality, compared to a gold standard protocol -involving only the lower limbs training- is more effective in improving ADL performance in terms of reduction of exercise time for a specific test (GLITTRE test). The secondary aims are to evaluate whether the combined training modality, compared to a gold standard protocol involving only the lower limbs, is more effective in a) increasing the effort tolerance of the lower limbs; b) increasing the effort tolerance of the upper limbs and c) reducing the energy cost of walking.

Methods:

This is a multicenter RCT study with a low-risk intervention.

Patients with a diagnosis of COPD, according to the Global Initiative for Lung Disease (GOLD) criteria, will be recruited for this purpose and randomly assigned to two groups: Lower limbs (LL) group and lower plus upper limbs (L+UL) group. The single list of randomization was created by a person external to the healthcare staff.

The treatment in the two groups is reported in the intervention section. All training sessions will be supervised by a physiotherapist. The initial training intensity both for lower and upper limbs will be determined on the basis of the load value performed in the last step of the maximal incremental effort test; the load value will be equal to 60% of the maximal wattage observed. Subsequently, the training intensity will be gradually increased during the sessions with a progression based on the symptoms, according to the protocol of Maltais et al. with steps of 10 watts for the lower limbs and 5 watts for the upper limbs.

During the rehabilitation period, formal education (alone or in groups) concerning the knowledge and management of the disease, healthy lifestyle, airway clearance, and inhaled drugs, will also be offered to all patients. Where indicated, airway clearance techniques and/or adaptation to non-invasive home ventilation will be administered.

At baseline, the investigators will collect clinical evaluations as follows:

* Demographic and anthropometric data
* Post-bronchodilator spirometry and plethysmography (Forced Expiratory Volume at 1 second, Forced Vital Capacity, Residual Volume, Inspiratory Capacity)
* Blood gas analysis in ambient air (PaO2, PaCO2, pH)
* Cumulative Illness Rating Score (CIRS)

Pre and post evaluations will be:

* Barthel Index
* EuroQoL

The Outcome measures are reported in the dedicated section.

The sample size has been calculated considering an improvement of the LL group of 23±20 seconds on the GLITTRE test corresponding to the MCID (Minimal Clinical Important Difference) for a standard GOLD rehabilitation treatment using a T-test for unpaired data with a= 0.05, b= 0.80. Estimating that patients in the L+UL group improve 22±20 seconds more than the LL group, the estimated sample is 30 patients (15 per group). Furthermore, considering a drop-out rate of 20%, it is estimated that 36 patients will be enrolled (12 patients per center).

The statistical evaluation will be conducted with the STATA 11 program (StataCorp LLC). Continuous variables will be expressed as mean and standard deviation (or median and quartiles) while categorical or binary variables as a percentage.

Statistical evaluation will be conducted with the use of appropriate parametric and non-parametric tests to verify differences between groups in treatment response (T-test or Wilcoxon to evaluate the difference between means or medians and chi-square test to evaluate the difference between frequencies). A secondary evaluation by logistic regression will also be performed to verify the baseline characteristics predictive of improvement in responders. A p value <.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* GOLD class 2-3 COPD
* Forced Expiratory Volume in the first second (FEV1) between 30% and 70% of the predicted value
* ability to walk and climb stairs without assistance
* stable clinical condition (pH > 7.35)

Exclusion Criteria:

* chronic respiratory insufficiency on long-term oxygen therapy (LTOT)
* severe orthopedic, neurological or cardiological comorbidities
* cognitive impairment
* recent exacerbation (within 15 days) requiring a change in therapy
* presence of lung disease other than COPD
* terminality

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in ADLs (GLITTRE test) | Time Frame. From the date of randomization to the End of the program (up to 16 days)
  To evaluate the improvement in terms of change of exercise time for a specific test (GLITTRE test)

SECONDARY OUTCOMES:
Change in effort tolerance of the lower limbs | Time Frame. From the date of randomization to the End of the program (up to 16 days)
  To evaluate the improvement in terms of change in the walked distance at 6 minutes walking test (6MWT)
Change in effort tolerance of the upper limbs | Time Frame. From the date of randomization to the End of the program (up to 16 days)
  To evaluate the improvement in terms of change in Tlim (time to exhaustion) in the Unsupported Upper Limb Exercise Test (UULEX)
Change in the energy cost of walking (EC) | Time Frame. From the date of randomization to the End of the program (up to 16 days)
  To evaluate the improvement in terms of change of the energy cost of walking with the EC test performed on a treadmill at a speed of 3.0 km/h for 6 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Michele Vitacca, MD, Study Director — ICS Maugeri IRCCS, respiratory rehabilitation of the Institute of Lumezzane
Locations (3):
- Italy (3):
  - ICS Maugeri IRCCS, Respiratory rehabilitation of the Institute of Lumezzane, Lumezzane, Brescia
  - ICS Maugeri IRCCS, Respiratory rehabilitation of the Institute of Montescano, Montescano, Pavia
  - ICS Maugeri IRCCS, Respiratory rehabilitation of the Institute of Tradate, Tradate, Varese

REFERENCES:
- [Background] Olopade CO, Beck KC, Viggiano RW, Staats BA. Exercise limitation and pulmonary rehabilitation in chronic obstructive pulmonary disease. Mayo Clin Proc. 1992 Feb;67(2):144-57. doi: 10.1016/s0025-6196(12)61316-0. PMID 1545579
- [Background] O'Donnell DE, Laveneziana P, Webb K, Neder JA. Chronic obstructive pulmonary disease: clinical integrative physiology. Clin Chest Med. 2014 Mar;35(1):51-69. doi: 10.1016/j.ccm.2013.09.008. Epub 2013 Dec 12. PMID 24507837
- [Background] Vaes AW, Wouters EFM, Franssen FME, Uszko-Lencer NHMK, Stakenborg KHP, Westra M, Meijer K, Schols AMWJ, Janssen PP, Spruit MA. Task-related oxygen uptake during domestic activities of daily life in patients with COPD and healthy elderly subjects. Chest. 2011 Oct;140(4):970-979. doi: 10.1378/chest.10-3005. Epub 2011 Mar 17. PMID 21415128
- [Background] Bendixen HJ, Waehrens EE, Wilcke JT, Sorensen LV. Self-reported quality of ADL task performance among patients with COPD exacerbations. Scand J Occup Ther. 2014 Jul;21(4):313-20. doi: 10.3109/11038128.2014.899621. Epub 2014 Mar 21. PMID 24649946
- [Background] van Helvoort HA, Willems LM, Dekhuijzen PR, van Hees HW, Heijdra YF. Respiratory constraints during activities in daily life and the impact on health status in patients with early-stage COPD: a cross-sectional study. NPJ Prim Care Respir Med. 2016 Oct 13;26:16054. doi: 10.1038/npjpcrm.2016.54. PMID 27734959
- [Background] Kapella MC, Larson JL, Covey MK, Alex CG. Functional performance in chronic obstructive pulmonary disease declines with time. Med Sci Sports Exerc. 2011 Feb;43(2):218-24. doi: 10.1249/MSS.0b013e3181eb6024. PMID 20543752
- [Background] Spruit MA, Singh SJ, Garvey C, ZuWallack R, Nici L, Rochester C, Hill K, Holland AE, Lareau SC, Man WD, Pitta F, Sewell L, Raskin J, Bourbeau J, Crouch R, Franssen FM, Casaburi R, Vercoulen JH, Vogiatzis I, Gosselink R, Clini EM, Effing TW, Maltais F, van der Palen J, Troosters T, Janssen DJ, Collins E, Garcia-Aymerich J, Brooks D, Fahy BF, Puhan MA, Hoogendoorn M, Garrod R, Schols AM, Carlin B, Benzo R, Meek P, Morgan M, Rutten-van Molken MP, Ries AL, Make B, Goldstein RS, Dowson CA, Brozek JL, Donner CF, Wouters EF; ATS/ERS Task Force on Pulmonary Rehabilitation. An official American Thoracic Society/European Respiratory Society statement: key concepts and advances in pulmonary rehabilitation. Am J Respir Crit Care Med. 2013 Oct 15;188(8):e13-64. doi: 10.1164/rccm.201309-1634ST. PMID 24127811
- [Background] Vaes AW, Delbressine JML, Mesquita R, Goertz YMJ, Janssen DJA, Nakken N, Franssen FME, Vanfleteren LEGW, Wouters EFM, Spruit MA. Impact of pulmonary rehabilitation on activities of daily living in patients with chronic obstructive pulmonary disease. J Appl Physiol (1985). 2019 Mar 1;126(3):607-615. doi: 10.1152/japplphysiol.00790.2018. Epub 2018 Nov 29. PMID 30496707
- [Background] Thomas MJ, Simpson J, Riley R, Grant E. The impact of home-based physiotherapy interventions on breathlessness during activities of daily living in severe COPD: a systematic review. Physiotherapy. 2010 Jun;96(2):108-19. doi: 10.1016/j.physio.2009.09.006. Epub 2010 Jan 18. PMID 20420957
- [Background] Marques A, Gabriel R, Jacome C, Cruz J, Brooks D, Figueiredo D. Development of a family-based pulmonary rehabilitation programme: an exploratory study. Disabil Rehabil. 2015;37(15):1340-6. doi: 10.3109/09638288.2014.964376. Epub 2014 Sep 25. PMID 25255297
- [Background] Larson JL, Covey MK, Wirtz SE, Berry JK, Alex CG, Langbein WE, Edwards L. Cycle ergometer and inspiratory muscle training in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1999 Aug;160(2):500-7. doi: 10.1164/ajrccm.160.2.9804067. PMID 10430720
- [Background] McKeough ZJ, Velloso M, Lima VP, Alison JA. Upper limb exercise training for COPD. Cochrane Database Syst Rev. 2016 Nov 15;11(11):CD011434. doi: 10.1002/14651858.CD011434.pub2. PMID 27846347
- [Background] Hopp L, Walker J. Effectiveness of arm exercise on dyspnea in patients with chronic obstructive pulmonary disease: a systematic review. JBI Libr Syst Rev. 2009;7(31):1353-1372. doi: 10.11124/01938924-200907310-00001. PMID 27820307
- [Background] Janaudis-Ferreira T, Hill K, Goldstein R, Wadell K, Brooks D. Arm exercise training in patients with chronic obstructive pulmonary disease: a systematic review. J Cardiopulm Rehabil Prev. 2009 Sep-Oct;29(5):277-83. doi: 10.1097/HCR.0b013e3181b4c8d0. PMID 19935139
- [Background] Kathiresan G, Jeyaraman SK, Jaganathan J. Effect of upper extremity exercise in people with COPD. J Thorac Dis. 2010 Dec;2(4):223-36. doi: 10.3978/j.issn.2072-1439.2010.11.4. PMID 22263051
- [Background] McKeough ZJ, Bye PT, Alison JA. Arm exercise training in chronic obstructive pulmonary disease: a randomised controlled trial. Chron Respir Dis. 2012 Aug;9(3):153-62. doi: 10.1177/1479972312440814. Epub 2012 Mar 27. PMID 22452973
- [Background] Clini E, Foglio K, Bianchi L, Porta R, Vitacca M, Ambrosino N. In-hospital short-term training program for patients with chronic airway obstruction. Chest. 2001 Nov;120(5):1500-5. doi: 10.1378/chest.120.5.1500. PMID 11713126
- [Background] Borg G. Perceived exertion as an indicator of somatic stress. Scand J Rehabil Med. 1970;2(2):92-8. No abstract available. PMID 5523831
- [Background] Maltais F, LeBlanc P, Jobin J, Berube C, Bruneau J, Carrier L, Breton MJ, Falardeau G, Belleau R. Intensity of training and physiologic adaptation in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 1997 Feb;155(2):555-61. doi: 10.1164/ajrccm.155.2.9032194.
- [Background] American Thoracic Society; American College of Chest Physicians. ATS/ACCP Statement on cardiopulmonary exercise testing. Am J Respir Crit Care Med. 2003 Jan 15;167(2):211-77. doi: 10.1164/rccm.167.2.211. No abstract available. PMID 12524257
- [Background] Gulart AA, Araujo CLP, Munari AB, Santos KD, Karloh M, Foscarini BG, Dal Lago P, Mayer AF. The minimal important difference for Glittre-ADL test in patients with chronic obstructive pulmonary disease. Braz J Phys Ther. 2020 Jan-Feb;24(1):54-60. doi: 10.1016/j.bjpt.2018.11.009. Epub 2018 Nov 20. PMID 30497829
- [Background] Takahashi T, Jenkins SC, Strauss GR, Watson CP, Lake FR. A new unsupported upper limb exercise test for patients with chronic obstructive pulmonary disease. J Cardiopulm Rehabil. 2003 Nov-Dec;23(6):430-7. doi: 10.1097/00008483-200311000-00007. PMID 14646791
- [Background] Holland AE, Spruit MA, Troosters T, Puhan MA, Pepin V, Saey D, McCormack MC, Carlin BW, Sciurba FC, Pitta F, Wanger J, MacIntyre N, Kaminsky DA, Culver BH, Revill SM, Hernandes NA, Andrianopoulos V, Camillo CA, Mitchell KE, Lee AL, Hill CJ, Singh SJ. An official European Respiratory Society/American Thoracic Society technical standard: field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1428-46. doi: 10.1183/09031936.00150314. Epub 2014 Oct 30. PMID 25359355
- [Background] Gaesser GA, Brooks GA. Muscular efficiency during steady-rate exercise: effects of speed and work rate. J Appl Physiol. 1975 Jun;38(6):1132-9. doi: 10.1152/jappl.1975.38.6.1132. PMID 1141128
- [Background] Karloh M, Araujo CL, Gulart AA, Reis CM, Steidle LJ, Mayer AF. The Glittre-ADL test reflects functional performance measured by physical activities of daily living in patients with chronic obstructive pulmonary disease. Braz J Phys Ther. 2016 Apr 8;20(3):223-30. doi: 10.1590/bjpt-rbf.2014.0155. PMID 27437713
- [Background] Balestroni G, Bertolotti G. [EuroQol-5D (EQ-5D): an instrument for measuring quality of life]. Monaldi Arch Chest Dis. 2012 Sep;78(3):155-9. doi: 10.4081/monaldi.2012.121. Italian. PMID 23614330
- [Background] Parshall MB, Schwartzstein RM, Adams L, Banzett RB, Manning HL, Bourbeau J, Calverley PM, Gift AG, Harver A, Lareau SC, Mahler DA, Meek PM, O'Donnell DE; American Thoracic Society Committee on Dyspnea. An official American Thoracic Society statement: update on the mechanisms, assessment, and management of dyspnea. Am J Respir Crit Care Med. 2012 Feb 15;185(4):435-52. doi: 10.1164/rccm.201111-2042ST. PMID 22336677
- [Background] Jones PW, Harding G, Berry P, Wiklund I, Chen WH, Kline Leidy N. Development and first validation of the COPD Assessment Test. Eur Respir J. 2009 Sep;34(3):648-54. doi: 10.1183/09031936.00102509. PMID 19720809
- [Background] Bestall JC, Paul EA, Garrod R, Garnham R, Jones PW, Wedzicha JA. Usefulness of the Medical Research Council (MRC) dyspnoea scale as a measure of disability in patients with chronic obstructive pulmonary disease. Thorax. 1999 Jul;54(7):581-6. doi: 10.1136/thx.54.7.581. PMID 10377201